CLINICAL TRIAL: NCT01911663
Title: The Effect of Korean Red Ginseng Supplementation on Glucose Control in Subjects With Impaired Fasting Glucose, Impaired Glucose Tolerance or Newly-diagnosed Type 2 Diabetes Mellitus
Brief Title: The Effect of Korean Red Ginseng Supplementation on Glucose Control
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KGC-CKJ-PC
Record Dates: First submitted 2013-07-26; First posted 2013-07-30 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- KRG (Experimental): 500 mg Korea red ginseng (KRG)
  Interventions: Dietary Supplement: KRG
- Placebo (Placebo Comparator): 500 mg placebo (corn starch)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: KRG — 500 mg Korea red ginseng (KRG)
  Arms: KRG
Dietary Supplement: Placebo — 500 mg placebo
  Arms: Placebo

SUMMARY:
This study is a randomized, double-blind, placebo-controlled clinical trial designed to evaluate the effect of Korean red ginseng supplementation on glucose control in subjects with impaired fasting glucose, impaired glucose tolerance or newly-diagnosed type 2 Diabetes Mellitus and to establish a clinical evidence on glucose control effect of KRG.

DETAILED DESCRIPTION:
Study participants, who were all aged between 20 and 70, were recruited from health checkup center at Ilsan hospital (Gyeonggi-do, Korea) and the advertisements in local newspaper. After the glucose screening test, subjects with IFG (100 mg/dL ≤ fasting blood glucose ≤ 125mg/dL), IGT (140mg/dL ≤ 2-h OGTT), or newly-diagnosed T2DM (fasting glucose ≥ 126 mg/dL) were enrolled in this study. Exclusion criteria that all selected patients met were: 1) Taking glucose-lowering medications or having insulin injections. 2) Chronic alcoholism or having an evidence or alcoholism. 3) Pregnant or in breast feeding. 4) Having chronic gastrointestinal disorders. 5) Showing signs of nutrient deficiency of malnutrition. 6) Patients with serious kidney problems. 7) Patients with serious liver problems. 8) Patients whose job could be a threat when hypoglycemia occurs. 9) Patients who have experienced the complications such as headache, insomnia, heart palpitations and raised blood pressure after eating red ginseng. 10) Other patients who were considered unsuitable for this study by the researchers

This study was designed for 12-week randomized, double-blinded, placebo-controlled trial. Sixty subjects were randomly assigned to receive placebo (corn starch) or 500 mg KRG. Both group consumed 10 capsules per day, three times daily after breakfast (3 capsules), lunch (3 capsules) and dinner (4 capsules), and it comes to total 5.0g daily. Red ginseng and placebo capsules were provided by the Korea Ginseng Cooperation (KGC, Daejeon, Korea).

Subjects met with the investigational team at four different time points: Screening (Week -1), randomization and treatment baseline (Week 0), treatment midpoint (Week 6), and treatment endpoint (Week 12). Daily intake by 24-hour recall method and physical activity were measured at baseline (Week 0), midpoint (Week 6), and endpoint (Week 12) of the treatment period. Compliance with study restrictions and capsule consumption was monitored via daily documentation by subjects on individualized study calendars and end-study count of returned capsules.

ELIGIBILITY:
Inclusion Criteria:

* subjects with IFG (100 mg/dL ≤ fasting blood glucose ≤ 125mg/dL), IGT (140mg/dL ≤ 2-h OGTT), or newly-diagnosed T2DM (fasting glucose ≥ 126 mg/dL) were enrolled in this study.

Exclusion Criteria:

* Exclusion criteria that all selected patients met were: 1) Taking glucose-lowering medications or having insulin injections. 2) Chronic alcoholism or having an evidence or alcoholism. 3) Pregnant or in breast feeding. 4) Having chronic gastrointestinal disorders. 5) Showing signs of nutrient deficiency of malnutrition. 6) Patients with serious kidney problems. 7) Patients with serious liver problems. 8) Patients whose job could be a threat when hypoglycemia occurs. 9) Patients who have experienced the complications such as headache, insomnia, heart palpitations and raised blood pressure after eating red ginseng. 10) Other patients

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-11; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
change from baseline in glucose | 12 week

SECONDARY OUTCOMES:
change from baseline in insulin | 12 week
change from baseline in C-peptide | 12 week

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratory of clinical Nutrigenetics/Nutrigenomic, Seoul, South Korea